CLINICAL TRIAL: NCT03852134
Title: Milking of the Cut-Cord During Resuscitation of Preterm Infants: A Randomized Controlled Trial (The MOCC Study)
Brief Title: Milking of the Cut-Cord During Resuscitation of Preterm Infants (The MOCC Study)
Acronym: MOCC
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: IWK Health Centre (Other)
Responsible Party: Principal Investigator, Walid El-Naggar, Principle Investigator, Associate Professor of Pediatrics, IWK Health Centre
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MOCC Study
Record Dates: First submitted 2018-04-30; First posted 2019-02-25 (Actual); Last update posted 2019-02-25 (Actual); Status verified 2019-02

CONDITIONS: Preterm Infant
Keywords: preterm infant; delayed cord clamping; cord milking; resuscitation
MeSH Terms: conditions — Premature Birth

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MOCC Group (Experimental): The OB provider will hold the baby at/below the placenta, provide warmth, stimulate the baby and suction the mouth/nose for 30 secs.S/He will then clamp and cut the cord about 5 cm from the the introitus (vaginal deliveries) or from the abdominal incision (C-Sections) before handing the baby with the long-cut cord to the neonatal team to resuscitate/ stabilize the baby. A member of the neonatal team will milk the long-cut cord slowly 1 time from the cut end toward the infant over 10 secs before clamping and cutting the cord 1-2 cm from the umbilical stump. The neonatal team will provide PPV to the baby (during the milking process) if the baby is not breathing. If the baby is breathing during the milking process the team will continue the stabilization as per standard NRP practice.
  Interventions: Procedure: MOCC Group
- DCC group (Active Comparator): The OB provider will hold the baby at or below the level of placenta, provide warmth, stimulate the baby to breathe and suction the mouth/nose if needed for the first 30 seconds.
  After these initial 30 seconds, if the baby is breathing then the obstetrician will continue DCC for a total of 60 seconds before clamping and cutting the cord close to the umbilicus and handing over the baby to the neonatal team for further stabilization as per standard NRP practice. If the baby is not breathing after the initial 30 seconds of DCC, then the OB provider will clamp and cut the cord close to the umbilicus and hand over the baby to the neonatal team to continue resuscitation of the baby as per the standard NRP guidelines.
  Interventions: Procedure: DCC Group

INTERVENTIONS:
Procedure: MOCC Group — After 30 seconds of DCC, the cord will be clamped and cut 5 cm from the introitus in vaginal delivery or abdominal incision in the case of cesarean section before passing the infant with the long umbilical cord segment to the pediatric provider who will milk the cord one time towards the baby during resuscitation.
  Other Names: Monitoring cerebral oxygenation by NIRS
  Arms: MOCC Group
Procedure: DCC Group — The OB provider will hold the baby at or below the level of placenta, provide warmth, stimulate the baby to breathe and suction the mouth/nose if needed for the first 30 seconds.
  After these initial 30 seconds, if the baby is breathing then the obstetrician will continue DCC for a total of 60 seconds before clamping and cutting the cord close to the umbilicus and handing over the baby to the neonatal team for further stabilization as per standard NRP practice. If the baby is not breathing after the initial 30 seconds of DCC, then the OB provider will clamp and cut the cord close to the umbilicus and hand over the baby to the neonatal team to continue resuscitation of the baby as per the standard NRP guidelines.
  Other Names: Monitoring cerebral oxygenation by NIRS
  Arms: DCC group

SUMMARY:
In this feasibility study, the investigators will randomize preterm infants born at <32 weeks gestation to either the standard practice of delayed cord clamping (DCC) for 30-60 seconds at birth or milking of the long-cut cord (MOCC) while providing resuscitation/stabilization to the infant. The main objectives of the trial are to assess the feasibility of the new approach (MOCC) and to compare the two groups regarding the hemoglobin levels on admission to NICU in addition to neonatal morbidity and mortality.

ELIGIBILITY:
Inclusion Criteria:

* Preterm infants <32 weeks' gestation

Exclusion Criteria:

* Clinical evidence of interrupted placental circulation (placental abruption or avulsed cord) or bleeding from placenta previa.
* Monochorionic twins or any higher order multiple pregnancy
* Major fetal congenital or chromosomal abnormality
* Documented fetal anemia or in utero red blood cell transfusion
* Intent to withhold or withdraw treatment of the infant

Max Age: 1 Minute | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 98 (Estimated)
Dates: Start 2019-02-07 (Actual); Primary Completion 2021-02-07 (Estimated); Study Completion 2023-07-31 (Estimated)

PRIMARY OUTCOMES:
Rate of compliance to the study intervention | Two years
  to investigate the adherence to the new approach of MOCC during resuscitation/ stabilization following 30 seconds of DCC in preterm infants.
Number of patients completing the study | Two years
  To evaluate the number of patients who are recruited and completed the study to estimate the sample size needed for the design of a large multi-centre RCT.
Number of adverse events associated with the MOCC intervention | Till the participants reach 2 year- corrected age (around 4.5 years)
  To investigate any adverse events that could be attributed to the MOCC intervention.

SECONDARY OUTCOMES:
Compare hemoglobin (Hgb) concentration | From date of randomization and assessed up to 24 hours of age
  to compare hemoglobin (Hgb) concentration on NICU admission in preterm infants <32 weeks' gestation who receive MOCC during resuscitation/stabilization following 30 seconds of DCC with those who receive DCC alone for 30-60 seconds at birth (standard practice-control group).

OTHER OUTCOMES:
Temperature stability | From randomization assessed up to 2 hours of age
  Temperature on admission to NICU
Need for advanced resuscitation at birth | From randomization assessed up to 2 hours of age
  Need for advanced resuscitation including intubation, chest compressions and/or medications
Inotropic support | From randomization assessed up to 72 hours of age
  Need for inotropic medication support
Volume expander | From randomization assessed up to 72 hours of age
  Assess the need for a volume expander (saline bolus or albumin bolus)
Cerebral oxygenation | From randomization assessed up to 72 hours of age
  Measure the cerebral oxygenation using NIRS
Blood transfusion | From randomization assessed up to 36 weeks corrected gestational age
  Assess the number of blood transfusions baby received from birth
Intraventricular hemorrhage (IVH) | From randomization assessed up to 36 weeks corrected age
  Assess the grade of IVH
Long-term outcomes | 24 Months Corrected age
  Long-term neurodevelopmental outcomes at 18-24 months of corrected age.

CONTACTS AND LOCATIONS:
Overall Officials: Walid El-Naggar, Principal Investigator — IWK Health Centre
Locations (1):
- IWK Health Centre, Halifax, Nova Scotia, Canada

IPD SHARING:
Plan to Share IPD: No
IPD will not be shared

REFERENCES:
- [Derived] El-Naggar W, Mitra S, Abeysekera J, Disher T, Woolcott C, Hatfield T, McMillan D, Dorling J. Milking of the Cut Cord During Stabilization of Infants Born Very Premature: A Randomized Controlled Trial. J Pediatr. 2025 Mar;278:114444. doi: 10.1016/j.jpeds.2024.114444. Epub 2024 Dec 24. PMID 39722339